CLINICAL TRIAL: NCT07066878
Title: Survival, Complications and Quality of Life in Patients Affected by Head and Neck Cancer: a Retrospective Analysis
Brief Title: This Protocol Focuses on the Factors That Influence Survival, the Development of Complications and the Quality of Life Based on the Treatment Received in the Group of Patients Suffering From Malignant Lesions of the Head and Neck
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Galli, Principal Investigator, IRCCS San Raffaele
Other Study IDs: RETRO-HN
Record Dates: First submitted 2025-06-21; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Oral cavity cancer patients
  Interventions: Procedure: treatment received in the group of patients suffering from malignant lesions of the head and neck.
- Oropharyngeal cancer patiens
  Interventions: Procedure: treatment received in the group of patients suffering from malignant lesions of the head and neck.
- Laryngeal/Hypopharyngeal cancer patients
  Interventions: Procedure: treatment received in the group of patients suffering from malignant lesions of the head and neck.
- Major salivary glands cancer patients
  Interventions: Procedure: treatment received in the group of patients suffering from malignant lesions of the head and neck.

INTERVENTIONS:
Procedure: treatment received in the group of patients suffering from malignant lesions of the head and neck. — This protocol focuses on a retrospective, single-center analysis, analyzing the factors that influence survival as the main objective, and secondarily the development of complications and the quality of life based on the treatment received in the group of patients suffering from malignant lesions of the head and neck.

SUMMARY:
This protocol focuses on a retrospective, single-center analysis, analyzing the factors that influence survival as the main objective, and secondarily the development of complications and the quality of life based on the treatment received in the group of patients suffering from malignant lesions of the head and neck.

DETAILED DESCRIPTION:
Head and neck cancers (HNCs) comprise a heterogeneous group of malignancies arising from the mucosal epithelium of the upper aerodigestive tract, including the oral cavity, pharynx (nasopharynx, oropharynx, and hypopharynx), and larynx. These tumors are predominantly squamous cell carcinomas (HNSCC), although salivary gland malignancies and other histologic subtypes such as neuroendocrine tumors or sarcomas are also included in this anatomical classification. Globally, HNCs account for nearly 900,000 new cases and over 400,000 deaths annually, representing a significant burden in both high- and low-income countries.

Over the past decades, improvements in diagnostic imaging (e.g., PET/CT, MRI), surgical techniques (including transoral robotic surgery [TORS] and transoral laser microsurgery [TLM]), radiotherapy modalities (e.g., intensity-modulated radiotherapy [IMRT]), and systemic therapies (platinum-based chemotherapy, targeted agents such as cetuximab, and, more recently, immune checkpoint inhibitors like nivolumab and pembrolizumab) have reshaped the therapeutic landscape. Nevertheless, survival outcomes remain highly variable and largely dependent on tumor site, T and N classification, extranodal extension (ENE), perineural and lymphovascular invasion, margin status, HPV status (particularly in oropharyngeal carcinomas), and patient-related factors such as age, performance status, and comorbidities.

For early-stage tumors (Stage I-II), single-modality treatment-typically surgery or radiotherapy-achieves excellent oncologic outcomes with 5-year overall survival (OS) rates ranging from 70% to 90%. In contrast, patients with locally advanced disease (Stage III-IVB), particularly with hypopharyngeal or advanced laryngeal tumors, face significantly worse prognoses, with 5-year OS rates often below 40%, despite aggressive multimodality treatment. A notable exception is HPV-positive oropharyngeal squamous cell carcinoma (OPSCC), which exhibits favorable biology and enhanced responsiveness to chemoradiation, leading to OS rates exceeding 80-90%, even in advanced stages.

Treatment planning must balance oncologic control with functional preservation. While surgical resection (with or without microvascular reconstruction) remains a mainstay for many subsites, organ-preservation protocols based on concurrent chemoradiotherapy are often preferred for tumors of the oropharynx, hypopharynx, and larynx, particularly in functionally critical areas. However, definitive chemoradiation is associated with substantial acute and late toxicities, including mucositis, dysphagia, xerostomia, aspiration, and long-term dependence on feeding tubes or tracheostomy, which may severely impact health-related quality of life (HRQoL).

In this context, robust comparative analyses of different treatment modalities-taking into account tumor subsite, stage, treatment-related morbidity, complications (e.g., graded by the Clavien-Dindo classification), and validated patient-reported outcome measures such as the EORTC QLQ-H&N35 and the FACT-H&N-are critical for guiding evidence-based, patient-centered care. Understanding the oncologic efficacy, complication profile, and quality of life outcomes across treatment strategies is essential to inform multidisciplinary decision-making and optimize long-term survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to provide informed consent for study participation
* Age 18 years or older
* Histological diagnosis of head and neck cancer (any site, any histology)
* Treatment (surgical and/or radiotherapy and/or medical) received at San Raffaele Hospital between January 2014 and January 2024
* Consent for use of personal data for scientific purposes

Exclusion Criteria:

* Age under 18 years
* No histological diagnosis of head and neck cancer
* Treatment not performed at San Raffaele Hospital (surgical and/or radiotherapy and/or medical)
* Lack of signed consent for use of personal data for scientific purposes
* Severe comorbidities interfering with study participation or treatment protocols
* Inability to understand or provide informed consent due to cognitive or psychiatric disorders
* Concurrent participation in another clinical trial that may interfere with study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who have been diagnosed with a malignant lesion of the head and neck district (specifically at the level of the oral cavity, oropharynx, larynx, hypopharynx or parotid gland) and underwent treatment with curative purpose (specifically the treatment may be surgical alone, surgical followed by radiotherapy treatment and possible chemotherapy, or radiotherapy, in possible association with chemotherapy in an upfront setting).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in Patients with Head and Neck Malignancies Treated with Curative Intent | 5 years
  To assess overall survival in patients with malignant lesions of the head and neck (oral cavity, oropharynx, hypopharynx, larynx) undergoing curative treatment. Treatment modalities include major oncological surgery (alone or followed by adjuvant radiotherapy ± chemotherapy), definitive radiotherapy, definitive chemoradiotherapy, or induction chemotherapy followed by surgery or radiotherapy.
  Time Frame: 5 years from treatment initiation
  Unit of Measure: Time (months)

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Related Complications Classified by Clavien-Dindo Scale | 5 years
  To evaluate postoperative and post-therapy complications related to surgery, radiotherapy, and chemotherapy. Complications include hemorrhage, wound dehiscence, pharyngocutaneous fistula, flap necrosis, radiodermatitis, xerostomia, mucositis, cytopenia, sepsis, and organ dysfunction.
  Classification: Clavien-Dindo Classification of Surgical Complications (Grade I to V; higher grades indicate more severe complications)
  Time Frame: Assessed short-term (≤30 days) and medium-term (up to 12 months) post-treatment, with overall follow-up to 5 years
  Unit of Measure: Clavien-Dindo Grade (Ordinal scale: Grade I [minor] to Grade V [death])

OTHER OUTCOMES:
Health-Related Quality of Life (HRQoL) Measured by EORTC QLQ-H&N35 | 5 years
  To assess quality of life domains affected by head and neck cancer treatment, including pain, swallowing, speech, social eating, and appearance.
  Instrument: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck 35 (EORTC QLQ-H&N35)
  Scale Range: Scores range from 0 to 100 for each domain/subscale. Higher scores indicate greater symptom severity or worse quality of life.
  Time Frame: Evaluated at baseline and multiple time points up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No